CLINICAL TRIAL: NCT00814294
Title: An 18-Week Randomized, Double-Blind, Multicenter, Comparator Study of Two Doses of Oral HDV-Insulin and Placebo With Background Metformin Treatment in Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Two Doses of Oral HDV-Insulin and Placebo With Background Metformin Treatment in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Diasome Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP 01-2007-03
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Diabetes
Keywords: Type 2
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1; Placebo (Placebo Comparator): Patients receive a sugar pill.
  Interventions: Drug: placebo
- 2; Oral Hepatic Directed Vesicles (HDV)-Insulin (U-5) (Experimental): Patients receive Oral HDV-Insulin (U-5).
  Interventions: Drug: Oral Hepatic Directed Vesicles (HDV)-Insulin (U-5)
- 3; Oral Hepatic Directed Vesicles (HDV)-Insulin (U-15) (Experimental): Patients receive Oral HDV-Insulin (U-15).
  Interventions: Drug: Oral Hepatic Directed Vesicles (HDV)-Insulin (U-15)

INTERVENTIONS:
Drug: placebo — placebo capsule,0 units, quater in die (QID) for 18 weeks
  Arms: 1; Placebo
Drug: Oral Hepatic Directed Vesicles (HDV)-Insulin (U-15) — Oral HDV-I Caps; 15 U; quater in die (QID) for 18 weeks.
  Arms: 3; Oral Hepatic Directed Vesicles (HDV)-Insulin (U-15)
Drug: Oral Hepatic Directed Vesicles (HDV)-Insulin (U-5) — Oral HDV-I; Caps; 5 U; quater in die (QID) for 18 weeks.
  Arms: 2; Oral Hepatic Directed Vesicles (HDV)-Insulin (U-5)

SUMMARY:
The primary objective of this trial is to compare the reduction in mean glycated hemoglobin levels (HbA1c) between 2 doses of oral HDV-I and placebo in type 2 diabetic patients on background metformin therapy at the end of 18 weeks of treatment.

The secondary objectives are:

* To evaluate the effects of oral HDV-I versus placebo on the 7-point glucose test, fasting plasma glucose (FPG), insulin, homeostasis model assessment of insulin resistance (HOMA-IR), homeostasis model assessment of β-cell function (HOMA-β), frequency of hypoglycemic events, body weight, and lipid levels; and
* To evaluate the safety and tolerability of oral HDV-I.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study with a washout/stabilization period of up to 12 weeks in duration and an 18-week double-blind treatment period. There will be a total of 8 visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years, inclusive;
* Diagnosis of type 2 diabetes mellitus;
* Fasting plasma glucose <=250 mg/dL;
* BMI <=45 kg/m2;
* HbA1c levels as follows at Screening:
* On a stable dose of metformin monotherapy with an HbA1c >=7.5% and <=9.5%;
* On metformin and 1 other OAD (excluding TZD, exenatide, or insulin) with an HbA1c >=6.8% and <=9.0%;
* Naïve to antidiabetic therapy or have not been on a stable dose of metformin monotherapy for <12 weeks with an HbA1c >=8.0% and <=10.5%;
* Understanding of the study procedures and agreement to participate in the study, giving written informed consent;
* Women may be enrolled if all of the following criteria (in addition to the above criteria) are met:
* They are not pregnant (women of childbearing potential must have a negative serum pregnancy test at Visit 1);
* They are not breast-feeding;
* They do not plan to become pregnant during the study; and
* They have had a hysterectomy or tubal ligation 6 months prior to the study, have been post-menopausal for 1 year, or will practice a method of birth control throughout the study.

Exclusion Criteria:

* History of type 1 diabetes and/or history of ketoacidosis;
* History of chronic (>2 months) use of insulin therapy or recent initiation of insulin use intended for chronic administration;
* Use of TZD (pioglitazone or rosiglitazone) or exenatide within 3 months prior to Screening;
* Use of prescription or over the counter weight loss agents within 1 month prior to Screening;
* Use of any lipid-altering, antihypertensive, and other chronic use medication not stable for 1 month prior to Screening;
* Use of any medication that may alter blood glucose analyses;
* Any serious disorder including cardiac, pulmonary, hepatic, uncontrolled endocrine/metabolic, hematologic/oncologic (within the last 5 years), neurologic, and psychiatric diseases that would interfere with the conduct of the study or interpretation of the data;
* Require regular use of medication that interferes with the oral absorption and/or metabolism of insulin or metformin;
* History of pancreatitis;
* History of acquired immune deficiency syndrome or human immunodeficiency virus;
* History of drug or alcohol abuse within the past 2 years;
* Hospitalization for any cause within 14 days prior to the study;
* History of an allergic or toxic response to oral HDV-I;
* Uncontrolled hypertension: systolic blood pressure >160 mmHg and diastolic blood pressure >95 mmHg;
* Triglycerides >400 mg/dL;
* Aspartate aminotransferase or alanine aminotransferase >2.5 times the upper limit of normal (ULN);
* Creatine phosphokinase >3 times the ULN;
* Patients on a weight loss program with ongoing weight loss, or starting an intensive exercise program within 4 weeks of starting the study;
* Use of any investigational drug within 30 days preceding the first dose of study medication; or
* Employment by the research center.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to compare the reduction in mean glycated hemoglobin levels (HbA1c) between 2 doses of oral HDV-I and placebo in type 2 diabetic patients on background metformin therapy at the end of 18 weeks of treatment. | 18 weeks

SECONDARY OUTCOMES:
To evaluate the effects of oral HDV-I versus placebo on the 7-point glucose test | 18 weeks
To evaluate the effects of oral HDV-I versus placebo on fasting plasma glucose (FPG) and insulin | 18 weeks
To evaluate the effects of oral HDV-I versus placebo on the homeostasis model assessment of insulin resistance (HOMA-IR)and homeostasis model assessment of β-cell function (HOMA-β) | 18 Weeks
To evaluate the effects of oral HDV-I versus placebo on frequency of hypoglycemic events, body weight, and lipid levels | 18 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Len Rosenberg, PhD, RPh, Study Director — Diasome Pharmaceuticals; David Orloff, MD, Study Director — Medpace, Inc.
Locations (38):
- United States (38):
  - Muscle Shoals, Alabama
  - Litchfield Park, Arizona
  - Tucson, Arizona
  - Concord, California
  - Paramount, California
  - Sacramento, California
  - San Mateo, California
  - Stockton, California
  - Valley Village, California
  - Walnut Creek, California
  - Chiefland, Florida
  - Fort Lauderdale, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Topeka, Kansas
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Brockton, Massachusetts
  - Picayune, Mississippi
  - Omaha, Nebraska
  - Staten Island, New York
  - Cincinnati, Ohio
  - Delaware, Ohio
  - Zanesville, Ohio
  - Beaver, Pennsylvania
  - Kingsport, Tennessee
  - Corpus Christi, Texas
  - El Paso, Texas
  - Houston, Texas
  - Hurst, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Manassas, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
  - Milwaukee, Wisconsin